CLINICAL TRIAL: NCT05680714
Title: Does the Improved Coordination of Care for Fall- and Fracture Prevention in Oslo Have Effect on the Rate of Hip Fractures, Need of Nursing Homes or Death?
Brief Title: Does the New Fall- and Fracture Prevention Initiative in Oslo Have Effect?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Oslo (Other); Oslo University Hospital (Other); Oslo Municipality (Other Government)
Responsible Party: Principal Investigator, Haakon Eduard Meyer, Principal Investigator, Senior Medical Officer, Professor in Epidemiology and Preventive Medicine, Norwegian Institute of Public Health
Other Study IDs: RCN296587; 296587 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2022-12-13; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Fall Injury; Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Needs Assessment; Patient Care Team; Checklist; House Calls; Deprescriptions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- FALLERS IN THE INTERVENTION BOROUGHS: Fallers 65+ years from the borough of Nordstrand from January 1. 2015 Fallers 65+ years from the borough of Østensjø from September 1. 2016
  Fall injury will be included as a time-varying exposure variable. The individuals are all registered as non-fallers until they are registered with a fall injury in the NPR database, when they shift status to fallers.
  Interventions: Other: Implement coordination of care with multifactorial falls- and fracture risk assessment and tailored intervention
- FALLERS IN THE CONTROL BOROUGHS: Fallers 65+ years from all the 13 other boroughs of Oslo.
  Fall injury will be included as a time-varying exposure variable. The individuals are all registered as non-fallers until they are registered with a fall injury in the NPR database, when they shift status to fallers.
- NON-FALLERS: All non-fallers 65+ years from all Oslo boroughs.

INTERVENTIONS:
Other: Implement coordination of care with multifactorial falls- and fracture risk assessment and tailored intervention
  Other Names: Needs assessment and user involvement; Casefinding with identifying high risk individuals; Single point of entry to care in the boroughs; Cross sectoral plan for follow-up with role clarification; Interdisciplinary teams; Tools for multifactorial falls and fracture risk assessment (checklists for GP, home visits, injury clinic, osteoporosis); Information sharing; Primary and specialist care referral pathways; Targeted interventions (Ex: exercise, home safety, osteoporosis treatment, deprescribing, medical assessment); Champions to create enthusiasm and carry the intervention forward; Collaborative education of health professionals; Technology enablers in the electronic patients records
  Groups: FALLERS IN THE INTERVENTION BOROUGHS

SUMMARY:
The goal of this controlled before and after study is to evaluate a new patient pathway for patients 65 years and older who have suffered a fall injury.

The main questions the study aims to answer are whether this preventive initiative with improved care coordination reduces risk of subsequent hip fractures, admittance to nursing homes or death.

Researchers will compare two boroughs in Oslo who implemented the new patient pathway with the 13 other boroughs who did not reorganize their follow-up, but continued their care as usual.

DETAILED DESCRIPTION:
The study is an evaluation of a new patient follow-up for fall prevention in Oslo with improvement of coordination of care for elderly at risk of fall injuries.

The intervention were introduced to the boroughs of Nordstrand and Østensjø, which are compared to the other 13 boroughs of Oslo in this controlled before and after study.

THE COHORT

All persons 65 years and older in Oslo are included in Oslo Fall Cohort and we follow all cohort participants prospectively.

OUTCOME VARIABLES

* Hip fracture
* Long term admittance to nursing home
* Death

TIMELINE

The investigators have defined the following dates as the start of intervention:

1. Start of intervention in Nordstrand borough is set to January 1, 2015.
2. Start of intervention Østensjø borough is set to September 1, 2016.

In the main analysis, fallers from the two intervention boroughs, Nordstrand and Østensjø, will be compared with fallers from the control boroughs during the intervention. Any differences between the intervention and control boroughs before the intervention started will be taken into account.

Data on all participants are available from 2010, and the participants will be followed from January 2012 until December 2019.

For each analysis, persons with a hip fracture or living in a nursing home at baseline will be excluded.

The analysis in the evaluation is based on registry data and no analysis relating the intervention to the outcomes has been done before registration in clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Living on Oslo, Norway in the period January 1. 2012 - December 31. 2019

Exclusion Criteria:

* Hip fracture before baseline
* Living in nursing home at baseline

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Total population in Oslo 65 years or older in the period 2012 - 2019.
Sampling Method: Probability Sample
Enrollment: 121000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Hip fracture | 2012-2019
  A new hip fracture registered in the Norwegian Patient registry
Admission to nursing home | 2012-2019
  Long-term admission to nursing home
Death | 2012-2019
  Total mortality

SECONDARY OUTCOMES:
Subsequent fall injuries | 2012-1019
  Subsequent falls that result in injuries registered in the Norwegian Patient Registry

CONTACTS AND LOCATIONS:
Overall Officials: Gro Idland, PhD, Study Director — Municipality of Oslo, Department of Health

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT05680714/Prot_SAP_000.pdf